CLINICAL TRIAL: NCT06039644
Title: To Evaluate the Efficacy of Probiotics in Improvement and Prevention of Chemotherapy Associated Side Effectes in Patients with the Breast Cancer
Brief Title: To Evaluate the Clinical Efficacy of Probiotics in Patients with the Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GenMont Biotech Incorporation (Industry)
Collaborators: Mackay Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BC2023
Record Dates: First submitted 2023-09-06; First posted 2023-09-15 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: probiotics; chemotherapy side-effects; Breast carcinoma; gut microbiot; Lactobacillus reuteri; Lactobacillus plantarum; Lactobacillus paracasei
MeSH Terms: conditions — Breast Neoplasms | interventions — Probiotics; Control Groups

STUDY DESIGN:
Intervention Model Description: Parallel Assignment, Randomized Controlled Trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic group (Experimental): Subjects received two probiotic sachets per day
  Interventions: Dietary Supplement: Probiotic
- Placebo group (Placebo Comparator): Subjects received two placebo sachets per day
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Three-strain probiotic supplement includes Lactobacillus reuteri GMNL-89 (alive), Lactobacillus plantarum GMNL-141 (alive) and Lactobacillus paracasei GMNL-133 (alive).
  Other Names: Test group
  Arms: Probiotic group
Other: Placebo — Same additives to Probiotic group but replace probiotics with corn starch and Maltodextrin.
  Other Names: Control group
  Arms: Placebo group

SUMMARY:
Chemotherapy-associated side-effects would affect therapeutic effect, quality of life, and cause permanent harm to breast cancer patients. This study is designed to explore after consumption of probiotics of lactobacillus composite strain powder sachets for 6 months in breast cancer chemotherapy, and whether the improvement of meliorate the side effects, further assists patients completing the chemotherapy.

DETAILED DESCRIPTION:
In 2020, the incidence rate of women's breast cancer in Taiwan was up to 82.1% . The death rate increased to 16%; in 2021, the ranking rose to no.3, and the death rate grew up to 24.6%. In the decades, breast cancer gradually becomes the dominant malignant women's cancer in Taiwan. Besides the lumpectomy, chemotherapy is one of the dominant and important treatments for breast cancer. Beyond the effects of chemotherapy, several side effects rise up. The most common chemotherapy are anthracyclin drugs (doxorubicin and epirubicin) and taxane (docetaxel and paclitaxel ). There are common side effects including neutropenia, hair loss, vomiting, diarrhea, stomatitis, mucositis, peripheral neuropathy, dermatitis, nephrotoxicity, and hepatotoxicity. Currently, most treatments for chemotherapy-induced side effects are symptomatic treatment, but there is no good solution to prevent it.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-III breast patients using anthracycline-based and taxane-based chemotherapy (not limited before or after chemotherapy/surgery)
* BMI > 18 kg/m^2
* Age between 20 and 80 years old
* Patients judged by physicians to participate in this trial and who are willing

Exclusion Criteria:

* Pregnant or lactating female patients
* Patients with bariatric surgery, gastrointestinal resections, Crohn's disease, celiac disease
* BMI < 18 kg/m^2
* Patient who have severe allergy to soybeans or peanuts
* Those who are under 20 years old or over 80 years old

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change from 12 weeks in the chemotherapy associated side-effects questionnaire at 24 weeks | 24 weeks
  The questionnaire will finished to record the side effects, including nausea, vomiting, diarrhea, stomatitis, peripheral neuropathy, skin rashes, and hand-food syndrome before and after the treatment.

SECONDARY OUTCOMES:
Change from 12 weeks in self-record of the FACT-G questionnaire (The Functional Assessment of Cancer Therapy - General; Version 4) at 24 weeks | 24 weeks
  The FACT-G questionnaire will record the quality of life by subjects at 12-weeks and-24 weeks. There are 4 domains of quality of life will be measured, including physical well-being, social/family well-being, emotional well-being, functional well-being. All domains will sum as total score of 108, and each domain will also evaluated.
Variability in BMI (Body Mass Index) | 24 weeks
  BMI will calculated with weight and height combined in kg/m^2. Measured every visit (week 0. 3. 6. 9. 12. 15. 18. 21. 24)
Change from baseline in levels of hs-CRP (high-sensitivity C-Reactive Protein) in mg/dL at 12 weeks | 12 weeks
  Blood samples will collected to examine the variation of hs-CRP from baseline at 12 weeks.
Change from baseline in levels of hs-CRP (high-sensitivity C-Reactive Protein) in mg/dL at 24 weeks | 24 weeks
  Blood samples will collected to examine the variation of hs-CRP from baseline at 24 weeks.
Change from baseline in levels of IL-6 (Interleukin-6) in pg/mL at 12 weeks | 12 weeks
  Blood samples will collected to examine the variation of IL-6 from baseline at 12 weeks.
Change from baseline in levels of IL-6 (Interleukin-6) in pg/mL at 24 weeks | 24 weeks
  Blood samples will collected to examine the variation of IL-6 from baseline at 24 weeks.
Change from baseline in levels of IL-10 (Interleukin-10) in pg/mL at 12 weeks | 12 weeks
  Blood samples will collected to examine the variation of IL-10 from baseline at 12 weeks.
Change from baseline in levels of IL-10 (Interleukin-10) in pg/mL at 24 weeks | 24 weeks
  Blood samples will collected to examine the variation of IL-10 from baseline at 24 weeks.
Change from baseline in levels of TNF-α (Tumor Necrosis Factor-α) in pg/mL at 12 weeks | 12 weeks
  Blood samples will collected to examine the variation of TNF-α from baseline at 12 weeks.
Change from baseline in levels of TNF-α (Tumor Necrosis Factor-α) in pg/mL at 24 weeks | 24 weeks
  Blood samples will collected to examine the variation of TNF-α from baseline at 24 weeks.
Change from baseline in gut microbiome at 12 weeks | 12 weeks
  Fecal sample will collected to extract DNA from the intestinal microbiota to examine the variations of gut microbiome from baseline at 12 weeks by NGS (Next Generation Sequencing) analysis.
Change from baseline in gut microbiome at 24 weeks | 24 weeks
  Fecal sample will collected to extract DNA from the intestinal microbiota to examine the variations of gut microbiome from baseline at 24 weeks by NGS (Next Generation Sequencing) analysis.
Variability in levels of ALT (Alanine Aminotransferase) in IU/L | 24 weeks
  ALT levels will obtained from routine medical records every visit. (week 0. 3. 6. 9. 12. 15. 18. 21. 24)
Variability in levels of AST (Aspartate Aminotransferase) in IU/L | 24 weeks
  AST levels will obtained from routine medical records every visit. (week 0. 3. 6. 9. 12. 15. 18. 21. 24)
Variability in levels of Creatinine in mg/dL | 24 weeks
  Creatinine levels will obtained from routine medical records every visit. (week 0. 3. 6. 9. 12. 15. 18. 21. 24)
Variability in levels of Hb (Hemoglobin) in g/dL | 24 weeks
  Hb levels will obtained from routine medical records every visit. (week 0. 3. 6. 9. 12. 15. 18. 21. 24)
Variability in levels of RBC (Red Blood Cell count) in 10^6/μL | 24 weeks
  RBC levels will obtained from routine medical records every visit. (week 0. 3. 6. 9. 12. 15. 18. 21. 24)
Variability in levels of Ht (Hematocrite) in % | 24 weeks
  Ht levels will obtained from routine medical records every visit. (week 0. 3. 6. 9. 12. 15. 18. 21. 24)
Variability in levels of WBC(White Blood Cell count) in 10^3/μL | 24 weeks
  WBC levels will obtained from routine medical records every visit. (week 0. 3. 6. 9. 12. 15. 18. 21. 24)
Variability in levels of MCV (Mean Corpuscular Volume) in fL | 24 weeks
  MCV levels will obtained from routine medical records every visit. (week 0. 3. 6. 9. 12. 15. 18. 21. 24)
Variability in levels of MCH (Mean Corpuscular Haemoglobin) in Pg | 24 weeks
  MCH levels will obtained from routine medical records every visit. (week 0. 3. 6. 9. 12. 15. 18. 21. 24)
Variability in levels of MCHC (Mean Corpuscular Haemoglobin Concentration) in g/dL | 24 weeks
  MCHC levels will obtained from routine medical records every visit. (week 0. 3. 6. 9. 12. 15. 18. 21. 24)
Variability in levels of ANC (Absolute Neutrophil Count) in mm^3 | 24 weeks
  Total neutrophils and WBC collected from routine medical records at each visit to calculate ANC levels. (week 0. 3. 6. 9. 12. 15. 18. 21. 24) ANC is calculated as 10 x WBC count in 1000s x (%Segment neutrophils + % bands neutrophils).
Variability in levels of platelet in 10^3/μL | 24 weeks
  Platelet levels will obtained from routine medical records every visit. (week 0. 3. 6. 9. 12. 15. 18. 21. 24)

CONTACTS AND LOCATIONS:
Overall Officials: Po-Sheng Yang, MD, PhD, Principal Investigator — Mackay Memorial Hospital
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No